CLINICAL TRIAL: NCT03385382
Title: Macular Thickness and Vessel Density Changes After Dexamethasone Implant and Ranibizumab Intravitreal Injection in Diabetic Macular Edema: 6-month Follow-up
Brief Title: Ranibizumab Versus Dexamethasone Implant in Diabetic Macular Edema
Acronym: LED
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, LISA TOTO, Researcher, G. d'Annunzio University
Other Study IDs: UChieti
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Ranibizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dexamethasone group: Patients with diabetic macular edema receiving dexamethasone
  Interventions: Drug: Dexamethasone intravitreal implant 0.7 mg
- ranibizumab: Patients with diabetic macular edema receiving ranibizumab
  Interventions: Drug: Ranibizumab Injection

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant 0.7 mg — Intravitreal Implant of dexamethasone
  Groups: Dexamethasone group
Drug: Ranibizumab Injection — Injection of ranibizumab
  Groups: ranibizumab

SUMMARY:
Between December 2016 and June 2017 a total of 40 eyes from 40 diabetic retinopathy patients with diabetic macular edema were recruited at the Ophthalmologic Clinic of University "G. d'Annunzio", Chieti-Pescara, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* BCVA greater than 0.5 LogMAR in the study eye at baseline examination
* Presence of recent DME
* CMT > 300µm as measured using the SD-OCT at the baseline examination

Exclusion Criteria:

* Any previous ocular surgery in the last 6 months
* Laser treatments
* Prior ocular trauma
* Retinal vascular diseases
* Vitreo-retinal interface diseases
* Medium lens opacities (according to Lens Opacities Classification System)

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with no proliferative moderate DR stage (simplified version of the ETDRS classification aimed by the American Academy of Ophthalmology Guidelines Committe) and cystoid macular edema type without subretinal fluid component were recruited
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | 6 months
  Decrease of macular thickness

SECONDARY OUTCOMES:
visual acuity | 6 months
  Increase of mean visual acuity

IPD SHARING:
Plan to Share IPD: No
Yes by request to the investigator via email